CLINICAL TRIAL: NCT00770276
Title: Mannheim Obesity Pilot Study: Evaluation of Metabolic Und Cardiovascular Risk in Obesity
Brief Title: Mannheim Obesity Study
Acronym: MOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Alexander Lammert, Dr. med., Universitätsmedizin Mannheim
Other Study IDs: MOS
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: obesity WHO I-III; metabolic syndrome; Framingham risk score; subclinical atherosclerosis; endothelial dysfunction
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bariatric surgery: Bariatric surgery
- conservative Therapie: diet and exercise

SUMMARY:
MOPS: Mannheim Obesity Pilot Study

Introduction:

Obesity is a central feature of the metabolic syndrome. With increasing prevalence of overweight and obesity, the incidence of WHO III° obesity will further augment. In this subset of obese patients, metabolic complications and cardiovascular risk are major clinical issues. Epidemiological data show that with increased BMI mortality rises (1). The SOS-Study demonstrated, for the first time, that bariatric surgery and consecutive weight reduction are associated with a decrease in cardiovascular and overall mortality. Significant mortality in this study was caused by cardiovascular events and cancer.

Metabolic Syndrome - MS - Despite varying definitions of the metabolic syndrome, obesity is one of its central features. Depending on the definition used, it can represent an obligate criterion (IDF) or a facultative parameter (WHO and ATP III). Even though not obligate, extreme obesity is a central risk factor for most other parameters of the metabolic syndrome.

Endothelial dysfunction -ED- represents the initial step of atherosclerosis (3). An appropriate measurement is the evaluation by retinal analysis. Epidemiological data demonstrate increased cardiovascular risk with retinal vessel pathology (4).

DETAILED DESCRIPTION:
Methods and procedures

Study design:

We conducted a prospective study in obesity WHO III° with consecutive enrollment. The study protocol was approved by the local ethics committee. Patients were recruited within an integrated concept designed for individuals seeking weight reduction. This network encompassed a complex approach by nutrition specialists, bariatric surgeons, endocrinologists, ENT specialists and psychologists. Patients could present themselves at any of the aforementioned specialists for study inclusion. Those who consented were followed, after conventional weight loss (diet, activity) or bariatric surgery 1 year later.

Evaluation:

Using a standardized form, we evaluated the medical and obesity history as well as associated metabolic complications (impaired glucose metabolism, elevated Cholesterol and NASH). We further inquired about regular medication, related diseases and classic cardiovascular risk factors (Framingham risk score: cardiovascular disease, family history of cardiovascular disease, nicotine abuse and arterial hypertension).

Anthropometry - Subsequently, a complete physical examination was conducted, taking into consideration the use of an adequate cuff to measure blood pressure. We further recorded circumferences of the neck, arm and waist (midway between the lower rib margin and iliac crest, with a measuring tape at the end of gentle expiration). Body weight and height were determined by calibrated scales to the nearest 0.1kg and cm, respectively.

Metabolism - Metabolic analysis was performed after an overnight fast. Baseline measurements included blood glucose, insulin, cholesterol, HDL, LDL, triglycerides and liver enzymes. Every individual without known diabetes was screened for the presence of impaired glucose metabolism by means of an OGTT. To exclude endocrine obesity we measured TSH levels and performed a one mg dexamethasone suppression test.

Intima media thickness (IMT) - Measurement of the intima media thickness of the right carotid artery was performed in order to detect subclinical vascular disease. Imaging protocol was executed according to the consensus statement of the American Society of Echocardiography (5).

Structural and functional endothelial dysfunction: Arterial and venous ratio (AVR) and flicker reaction - DVA was used for digital fundus imaging as well as conventional fundus examinations and retinal vessel analysis (RVA, imedos, Jena, Germany). Structural endothelial dysfunction was determined by arterial-venous ratio (AVR). After mydriasis with phenylephrine 10% and tropicamide 1%, images centred on the macula, the inferior arcade and the optic disc were recorded in both eyes. AVR was calculated by software after marking arteries and veins within two diameters of the optic disc (RVA, imedos, Jena, Germany).

Functional endothelial dysfunction was measured by flicker reaction of retinal vessels. This technique records dilatation of retinal vessels during and after exposure to flickering light. We used 1.5 mm segments of vessels within two disc diameters, which showed no crossing or bifurcation, and had a tortuosity < 30°. After baseline calibration, flickering light was shown for 20 seconds via interruption of continuous light at 12.5 Hz. During this period and for further 80 seconds, vessel diameter was continuously measured. To achieve higher reliability, this procedure was performed three times. Flicker of the artery and vein was expressed as the maximum in percent of the baseline diameter. Adjustment for eye movement was performed automatically by software. Details of this technique were published elsewhere (6-7).

BIA - Body composition was determined preoperatively by BIA. All patients were required to rest for 30 minutes, after which BIA was performed by applying 4 silver electrodes, with 2 detecting electrodes placed at the ulnar aspect of the right wrist and the right medial malleolus. After connecting the electrodes to the multiple-frequency BIA instrument (BIA 2000, Data Input, Darmstadt, Germany), measurements were recorded in real time via computer. The calculations for BCM, ECM, ECM/BCM, fat and TBW were performed using Nutri 2000 software (Data Input, Darmstadt, Germany).

Endpoints - The endpoint of our study was the identification of cardiovascular risk and metabolic complications or factors representing these risks in a population with obesity WHO. Therefore, we measured parameters of the metabolic syndrome, endothelial dysfunction and subclinical atherosclerosis. Patients, who gave informed consent, are followed after conventional weight loss (diet, activity) or bariatric surgery yearly. The decision for the type of intervention is connected to a complex process. According to the German obesity society subjects with more than 40 kg/m2 and patients with a BMI > 35 kg/m2 with obesity associated disease have the indication for bariatric surgery. After drafting of an expert's opinion for coverage of the costs by the health insurance patients may attend bariatric surgery. Because of the noncommittal character of the guideline of the German obesity society to health insurances not all patients will be able to get coverage for their surgery costs. Patients who are not able to get cost coverage or refuse surgery represent the conservative treatment (activity, diet). The interventional group will be treated by bariatric surgery (sleeve gastrectomy, Roux-en-Y gastric bypass). Therefore, the study has observational character.

ELIGIBILITY:
Inclusion Criteria:

* obesity WHO I-III

Exclusion Criteria:

* pregnancy
* acute vascular event within the last 3 months

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient department of an university hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2005-01; Primary Completion 2018-02 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome | baseline, after 1 and 2 years
Framingham risk score | baseline, 1 and 2 years
Subclinical atherosclerosis (IMT) | baseline, 1 and 2 years
Endothelial dysfunction | baseline, 1 and 2 years

SECONDARY OUTCOMES:
Change in body weight | baseline, 1 and 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Mannheim, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Calle EE, Thun MJ, Petrelli JM, Rodriguez C, Heath CW Jr. Body-mass index and mortality in a prospective cohort of U.S. adults. N Engl J Med. 1999 Oct 7;341(15):1097-105. doi: 10.1056/NEJM199910073411501. PMID 10511607
- [Background] Burguera B, Agusti A, Arner P, Baltasar A, Barbe F, Barcelo A, Breton I, Cabanes T, Casanueva FF, Couce ME, Dieguez C, Fiol M, Fernandez Real JM, Formiguera X, Fruhbeck G, Garcia Romero M, Garcia Sanz M, Ghigo E, Gomis R, Higa K, Ibarra O, Lacy A, Larrad A, Masmiquel L, Moize V, Moreno B, Moreiro J, Ricart W, Riesco M, Salinas R, Salvador J, Pi-Sunyer FX, Scopinaro N, Sjostrom L, Pagan A, Pereg V, Sanchez Pernaute A, Torres A, Urgeles JR, Vidal-Puig A, Vidal J, Vila M. Critical assessment of the current guidelines for the management and treatment of morbidly obese patients. J Endocrinol Invest. 2007 Nov;30(10):844-52. doi: 10.1007/BF03349226. PMID 18075287
- [Background] Davignon J, Ganz P. Role of endothelial dysfunction in atherosclerosis. Circulation. 2004 Jun 15;109(23 Suppl 1):III27-32. doi: 10.1161/01.CIR.0000131515.03336.f8. PMID 15198963
- [Background] Witt N, Wong TY, Hughes AD, Chaturvedi N, Klein BE, Evans R, McNamara M, Thom SA, Klein R. Abnormalities of retinal microvascular structure and risk of mortality from ischemic heart disease and stroke. Hypertension. 2006 May;47(5):975-81. doi: 10.1161/01.HYP.0000216717.72048.6c. Epub 2006 Apr 3. PMID 16585415
- [Background] Stein JH, Korcarz CE, Hurst RT, Lonn E, Kendall CB, Mohler ER, Najjar SS, Rembold CM, Post WS; American Society of Echocardiography Carotid Intima-Media Thickness Task Force. Use of carotid ultrasound to identify subclinical vascular disease and evaluate cardiovascular disease risk: a consensus statement from the American Society of Echocardiography Carotid Intima-Media Thickness Task Force. Endorsed by the Society for Vascular Medicine. J Am Soc Echocardiogr. 2008 Feb;21(2):93-111; quiz 189-90. doi: 10.1016/j.echo.2007.11.011. No abstract available. PMID 18261694
- [Background] Blum M, Bachmann K, Pietscher S, Brauer-Burchardt C, Vilser W, Strobel J. [Online measurement of retinal artery branches in type II diabetic patients. Initial clinical trials before and after laser coagulation]. Ophthalmologe. 1997 Oct;94(10):724-7. doi: 10.1007/s003470050193. German. PMID 9432241
- [Background] Blum M, Bachmann K, Wintzer D, Riemer T, Vilser W, Strobel J. Noninvasive measurement of the Bayliss effect in retinal autoregulation. Graefes Arch Clin Exp Ophthalmol. 1999 Apr;237(4):296-300. doi: 10.1007/s004170050236. PMID 10208262
- [Result] Lammert A, Hasenberg T, Kraupner C, Schnulle P, Hammes HP. Improved arteriole-to-venule ratio of retinal vessels resulting from bariatric surgery. Obesity (Silver Spring). 2012 Nov;20(11):2262-7. doi: 10.1038/oby.2012.122. Epub 2012 May 4. PMID 22555362
- [Result] Lammert A, Hasenberg T, Imhof I, Schnulle P, Benck U, Kramer BK, Hammes HP. High prevalence of retinal endothelial dysfunction in obesity WHO class III. Microvasc Res. 2012 Nov;84(3):362-6. doi: 10.1016/j.mvr.2012.09.004. Epub 2012 Sep 23. PMID 23009954
- [Derived] Mattern J, Lammert A, Otto M, Hammes HP. Retinopathy in an obesity WHO III cohort: prevalence and risk factors. Br J Ophthalmol. 2017 Nov;101(11):1550-1554. doi: 10.1136/bjophthalmol-2016-309566. Epub 2017 Mar 17. PMID 28314833
- [Derived] Lammert A, Nittka S, Otto M, Schneider-Lindner V, Kemmer A, Kramer BK, Birck R, Hammes HP, Benck U. Performance of the 1 mg dexamethasone suppression test in patients with severe obesity. Obesity (Silver Spring). 2016 Apr;24(4):850-5. doi: 10.1002/oby.21442. Epub 2016 Mar 7. PMID 26948683
- [Derived] Bachmayer C, Lammert A, Hasenberg T, Hammes HP. Healthy obese and post bariatric patients - metabolic and vascular patterns. Exp Clin Endocrinol Diabetes. 2013 Aug;121(8):483-7. doi: 10.1055/s-0033-1347248. Epub 2013 Jun 13. PMID 23765752